CLINICAL TRIAL: NCT02140996
Title: Ad-sig-hMUC-1/ecdCD40L Vector Vaccine for Immunotherapy of Epithelial Cancers
Brief Title: Safety Study of Human MUC-1 (Mucin-1) Adenoviral Vector Vaccine for Immunotherapy of Epithelial Cancers
Acronym: MUC-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Clinical Research Institute (Other)
Collaborators: MicroVAX, LLC (Unknown); ClinDatrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUC-1
Record Dates: First submitted 2014-05-08; First posted 2014-05-16 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Epithelial Cancers of the Lung, Breast, Ovary, Prostate and Colon
Keywords: MUC-1 vector vaccine; epithelial cancers; immunotherapy; safety; antigen specific vaccine, dendritic cell activation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad-sig-hMUC-1/ecdCD40L vector vaccine (Experimental): Experimental: Ad-sig-hMUC-1/ecdCD40L vector vaccine This trial has six cohorts with 3 subjects planned for each cohort. Subjects in the 1st cohort will receive 1 dose of vaccine injection at the lowest planned dose of the vector, 1 x 10^9 VP. If none of the patients in the 1st cohort experience Dose limiting toxicity (DLT), a 2nd cohort will receive 1 dose of 1x10^10 VP. If none of the patients in the 2nd cohort experience DLT, the dose escalation will continue with the 3rd cohort receiving 1 doses of 5 x 10^10 VP per injection. The patients in the 4th cohort will receive 1 injection of 1x10^11 if no DLT occurs in the preceding cohort. Additional patients will be added to cohort 5 or 6 if DLTs are encountered in the first 3 patients tested in each of these cohorts.
  Interventions: Drug: Ad-sig-hMUC-1/ecdCD40L vector vaccine

INTERVENTIONS:
Drug: Ad-sig-hMUC-1/ecdCD40L vector vaccine

SUMMARY:
In epithelial cancer, MUC-1(mucin-1) overexpression is thought to disrupt E-cadherin function, leading to anchorage-independent tumor cell growth and metastases. Elevated levels of MUC-1 expression have been found in patients with epithelial cancers of breast, ovarian, colon and lung. Furthermore, overexpression of MUC-1 is independently correlated with adverse clinical phenotypes, metastases and resistance to chemotherapy. In animal models, suppressing the expression of MUC-1 reduces the rates of growth and metastasis and increases the sensitivity of the cancer to chemotherapy-induced cell death.

In this study, an adenoviral Ad-sig-hMUC-1/ecdCD40L vector encoding a fusion protein in which the hMUC-1 epithelial antigen is attached to the CD40L (CD40 ligand). The preclinical results have also shown that two subcutaneous Ad-sig-hMUC-1/ecdCD40L vector injections can induce immunity through activation of dendritic cells and promotion of antigen specific B cells or antigen specific CD8 effector T cells which suppresses the growth of hMUC-1 tumor cells in 100% of the vaccinated mice without Interleukin (IL) 2 stimulation being required, this suggests that the Ad-sig-hMUC-1/ecdCD40L vector prime-hMUC-1/ecdCD40L protein boost has the potential to be an effective vaccine in epithelial tumors. Therefore, the safety and tolerability of the Ad-sig-hMUC-1/ecdCD40L vector vaccine will be tested in this phase I non-randomized open label dose escalation trial for men or women with metastatic or recurrent epithelial cancers of the lung, breast, ovary, prostate and colon.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women age 21 yrs or older with biopsy-proven recurrent or metastatic, measurable or non-measurable adenocarcinoma of the breast, ovary, lung, colon or prostate.
2. Elevated serum MUC-1 levels [as measured by Carcinoma Antigen (CA) 15-3 or CA27.29] at any time since the diagnosis of cancer (levels do not need to be elevated at the time of trial entry).
3. Received at least one line of palliative chemotherapy.
4. No chemotherapy and/or radiation therapy for at least 28 days before consent.
5. An echocardiogram that shows a left ventricular ejection fraction greater than or equal to the lower limits of normal.
6. Electrocardiogram (ECG) with no evidence of ischemia or infarction.
7. Ability to understand the study's risks, benefits, and procedures and provide written informed consent.
8. Performance status <2 on the Eastern Cooperative Oncology Group (ECOG) performance scale and life expectancy of greater than 12 months.
9. Acceptable pulmonary function. (If questionable a pulmonary function test will be performed.)
10. Negative serology for hepatitis B [hepatitis B surface antigen (HBsAg) negative], hepatitis C and human immunodeficiency virus (HIV).
11. All of the following: white blood count >3500, absolute neutrophil count >/= 1,500, hemoglobin > 8 g/dL, platelet count > 100,000/dL: Bilirubin <1.5, AST (aspartate aminotransferase), ALT (alanine aminotransferase), LDH (Lactate dehydrogenase) < 2 times the upper limit of normal, and calculated creatinine clearance >/= 50 mls/min.
12. For women with child-bearing potential: negative urinary pregnancy test at screening and within 7 days of enrollment; for men or women: willingness to use an approved contraceptive method while participating in this trial. Documentation of type of contraception patient will be using must be included in screening visit note by investigator.

Exclusion Criteria:

1. History of bronchospasm or asthma that requires steroid treatment (inhaled or oral).
2. Treatment with steroid (for any condition, except for chemotherapy premedication or emesis) within 28 days of trial registration.
3. Current anti-cancer treatment with doxorubicin (Adriamycin), lapatinib, trastuzumab, bevacizumab or other monoclonal antibody therapy. Patients must be off these therapies for at least 28 days. Patients may have been exposed to chemotherapy or radiation therapy 4 weeks prior to receiving the vaccination.
4. Current anti-cancer treatment with tamoxifen. Patients must be off tamoxifen for at least 28 days prior to enrollment. (Aromatase inhibitors and raloxifene are allowed).
5. History of any autoimmune disease such as lupus, rheumatoid arthritis or psoriasis.
6. Uncontrolled diabetes mellitus.
7. Unable or unwilling to undergo repeated clinical evaluations and other diagnostic procedures or unable to sign an informed consent.
8. History of other malignancies except squamous or basal cell carcinomas of the skin or cervical carcinoma in situ.
9. History of organ transplant or allogeneic bone marrow transplants.
10. Pregnant or nursing females.
11. Any acute or chronic viral, bacterial, or fungal infection which requires specific therapy. Acute therapy must be completed within 14 days prior to study treatment.
12. Any underlying conditions which would contraindicate therapy with study treatment (or allergies to reagents used in the study treatment).
13. Any history of cardiac disease including arrhythmia (requiring active treatment or medications), heart failure, angina, infarction or coronary artery disease.
14. History of hypercoagulable disorder including history of prior pulmonary embolism, antiphospholipid antibody syndrome, deep venous thrombosis [except for indwelling intravenous catheter associated DVT (deep vein thrombosis), as long as patient has completed anticoagulation therapy].
15. Any brain or leptomeningeal involvement by the cancer.
16. Known Ornithine transcarbamylase deficiency.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of a safe, tolerable, and immunologically active dose level of the Ad-sig-hMUC-1/ecdCD40L vector vaccine | Subjects will be followed up to 12 weeks after vaccine injection.
  Traditional 3+3 dose escalation scheme is employed for this trial. This trial has 6 cohorts with 3 subjects for each cohort. Subjects in the 1st cohort will receive the lowest planned dose of the vector, 1 x 10^9 VP. If no patient in the 1st cohort experiences Dose limiting toxicity (DLT), a 2nd cohort will receive 1 dose of 1x10^10 VP. Similarly, if no DLT occurs in the preceding cohorts, the dose escalation will continue with the 3rd cohort receiving 1 dose of 5 x 10^10 VP and the 4th cohort receiving 1 dose of 1x10^11 VP. Following completion of the 4th cohort, the toxicity of adding 1 or 2 booster injections at 7 and 21 days following the 1st vector injection will be tested in the 5th and 6th cohorts. The dose of each of the 2 or 3 vector injections administered in the 5th and 6th cohorts will be the top dose tolerated in the first 4th cohorts. If DLT is encountered in the first 3 patients in cohorts 5 or 6, then additional patients will be added to each of these cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Han Chong Toh, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - National Cancer Centre, Singapore